CLINICAL TRIAL: NCT00430196
Title: Placebo-Controlled Trial of BOTOX® Versus Zanaflex® for the Treatment of Subjects With Post Stroke Upper Limb Spasticity
Brief Title: BOTOX® Versus Zanaflex® for the Treatment of Post-Stroke or Traumatic Brain Injury Upper Limb Spasticity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO # 02-0510
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2007-01

CONDITIONS: Upper Limb Spasticity
MeSH Terms: interventions — Botulinum Toxins, Type A; tizanidine

INTERVENTIONS:
Drug: BOTOX®
Drug: Zanaflex®

SUMMARY:
In this study, we will compare BOTOX® versus Zanaflex ® for the treatment of muscle overactivity in the upper limb following stroke or brain traums. This is a critical step in the development of local intramuscular treatment for patients with muscle overactivity following an acute brain lesions, as opposed to the more classic oral treatments.

This study will be a multicenter, randomized, prospective, parallel, double blind study that enrolls subjects at twelve sites (including Mt. Sinai) throughout the United States and Europe. The purpose of this study is to evaluate the safety and efficacy of BOTOX® compared to Zanaflex® in reducing upper limb muscle tone in post-stroke subjects, as well as evaluating changes in muscle tone-related disability and drug-therapy tolerance. This will be an 18 week study. Subjects are eligible if they have been medically stable with upper limb spasticity 6 months after their first stroke. Subjects will be randomized to one of three treatment groups: Treatment Group I - intramuscular BOTOX® plus oral placebo, Treatment Group II - intramuscular placebo plus oral Zanaflex®, Treatment Group III - intramuscular placebo plus oral placebo. The dose of BOTOX® will be at the discretion of the investigator with a maximum of 500 U per subject. The dose of the Zanaflex® will be 4mg/day to a maximum of 36mg/day. The study anticipates that 150 subjects will be enrolled to provide sufficient information to answer the primary objective of safety and efficacy of the study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male and female subjects, of any race, between 18 and 85 years of age.
* Female subjects of childbearing potential must have a negative urine pregnancy test result at Visit 1/Screening. (A female is considered of childbearing potential unless she is postmenopausal or without a uterus and/or both ovaries.)
* Subjects with a history of stroke or traumatic brain injury, more than 90 days prior to Visit 2/Baseline, that result in disability caused by focal upper limb muscle over activity, as assessed by the Investigator and characterized by the following:

  * A wrist Ashworth tone of +3 or greater as measured on the Modified Ashworth Scale at Visit 1/Screening and Visit 2/Baseline;
  * A minimum measurement of +2 on the Disability Assessment Scale (DAS) for the principal therapeutic intervention target assessment (hygiene, dressing, pain, and cosmesis) chosen by the Investigator and the subject or subject's caregiver at Visit 1/Screening and Visit 2/baseline.
* Subjects, who, as assessed by the Investigator, clearly understand the intent of the study and are willing and able to comply with study instructions, complete the entire study and sign Informed Consent Form.

Exclusion Criteria:

* Female subjects who are pregnant (positive urine pregnancy test at Visit 1/screening), nursing, planning a pregnancy during the study period or female subjects of childbearing potential who are not using a reliable means of contraception. Reliable means of contraception. Reliable methods of contraception are hormonal methods or intrauterine device in use at least 14 days before study drug administration.
* Subjects with a severe contracture at the wrist (inability to passively move the joint more than 10 degrees) or a history of tendon transfer in the study limb.
* Subjects who have had a cast of the study limb within two weeks of the Visit 1/Screening or are planning casting of the study limb during the study period.
* Subjects with a diagnosis of Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis or any other disease that might interfere with neuromuscular function.
* Subjects with profound atrophy (as per the Investigator's assessment) of the muscle in the target area(s) of injection.
* Subjects with an infection at the injection site or systemic infection (in this case, postpone study entry until one week following recovery).
* Subjects with diagnosed orthostatic hypotension or subjects that are taking alpha-2 adrenergic agonists (e.g. clonidine).
* Subjects with impaired renal and/or hepatic function.
* Subjects with a known allergy or sensitivity to the study medications or its components.
* Subjects who are currently taking tizanidine or have taken tizandidine within 14 days prior to Visit 2/Baseline.
* Subjects who have received previous botulinum toxin injection(s) of any serotype into the target limb within 4 months of Visit 2/Baseline.
* Subjects who have received phenol or alcohol injections to the study limb.
* Subjects who are currently taking oral gabaergic medications (baclofen, gabapentin, benzodiazepines) or dantrolone sodium, or have been taking these drugs within 2 weeks of baseline (Visit 2). Please note that benzodiazepines will be excluded only as antispasmodic medications but not as hypnotics or anxiolytics on a PRN basis.
* Subjects who have not been on stable doses of their CNS medications (antidepressant, antianxiety drugs) for at least 2 months prior to Visit 1 (dose regimen must remain stable throughout the study).
* Subjects who are currently using medication that are contraindicated with the concomitant use of BOTOX® or Zanaflex®.
* Subjects currently participating in an investigational drug study or who have participated in an investigational drug study within 30 days of Visit 1/Screening.
* Subjects that in the Investigator's opinion have a concurrent condition that may put them at significant risk, may confound the study results, or may interfere significantly with the conduct of the study.
* Subjects with a history of poor cooperation, non-compliance with medical treatment, or unreliability.
* Subjects currently receiving anticoagulant therapy and who have an INR > 3.5

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135
Dates: Start 2003-12; Study Completion 2006-09

PRIMARY OUTCOMES:
wrist Modified Ashworth Score

SECONDARY OUTCOMES:
Disability Assessment Scale
Modified Frenchay Assessment
Walking Speed
Contralateral Grip Strength
Contralateral Finger Tap
Epworth Sleepiness Scale
Cognitive Evaluations Questionnaire
Discontinuation
Titration schedule of oral study medication between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: David Simpson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

REFERENCES:
- [Derived] Simpson DM, Gracies JM, Yablon SA, Barbano R, Brashear A; BoNT/TZD Study Team. Botulinum neurotoxin versus tizanidine in upper limb spasticity: a placebo-controlled study. J Neurol Neurosurg Psychiatry. 2009 Apr;80(4):380-5. doi: 10.1136/jnnp.2008.159657. Epub 2008 Oct 31. PMID 18977811